CLINICAL TRIAL: NCT01210053
Title: This Phase II Trial is Studying Sunitinib to See How Well it Works When Given as Maintenance Therapy in Treating Patients With Stage III or Stage IV Non-small Cell Lung Cancer Which is Previously Treated With Combination Chemotherapy.
Brief Title: Sunitinib as Maintenance Therapy in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: yangzhenzhou, Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yang-001
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Patients receive oral sunitinib malate 25 mg daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: malate Given orally

INTERVENTIONS:
Drug: malate Given orally — Patients receive oral sunitinib malate 25 mg daily in the absence of disease progression or unacceptable toxicity.
  Other Names: sutent

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether sunitinib is effective in treating non-small cell lung cancer.

PURPOSE: This phase II trial is studying sunitinib to see how well it works when given as maintenance therapy in treating patients with stage III or stage IV non-small cell lung cancer which is previously treated with combination chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the effect of sunitinib malate on the progression-free survival of patients with stage IIIB or IV non-small cell lung cancer Secondary
* To evaluate the toxicity of sunitinib when administered in the maintenance setting.
* To evaluate the additional response rate to sunitinib malate when administered in the maintenance setting.
* To evaluate the overall survival of patients treated with sunitinib. After completion of study treatment, patients are followed every 2 months for 1 year, every 6 months for 1 year, and periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* No evidence of symptomatic or untreated brain metastases, spinal cord compression, or carcinomatous meningitis
* Histologically or cytologically confirmed primary non-small cell lung cancer who have stable or responding disease after prior treatment with 3-6 courses of platinum -based therapy
* Not a candidate for combined modality therapy
* No cavitary lesions

Exclusion Criteria:

* Evidence of symptomatic or untreated brain metastases, spinal cord compression, or carcinomatous meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-11 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years

SECONDARY OUTCOMES:
• Grade and type of toxicity • 1-year survival rate • Response rate • Overall survival • Grade and type of toxicity • 1-year survival rate • Response rate • Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: yang zhenzhou, doctor, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China